CLINICAL TRIAL: NCT03286738
Title: Pattern of Use of Bevacizumab or Cetuximab in Patients With Metastatic Colorectal Cancer When Added to FOLFIRI Regimen as First-line Treatment; Multicenter, Registry Study
Brief Title: Pattern of Use of Bevacizumab or Cetuximab + FOLFIRI Regimen as First-line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joong Bae Ahn (Other)
Responsible Party: Sponsor-Investigator, Joong Bae Ahn, Professor, Yonsei University
Organization: Yonsei University (Other)
Other Study IDs: CTP_401
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FOLFIRI, target agent — * Irinotecan (Camtop Injection®, CJ HealthCare Corp.), Leucovorin, 5-Fluorouracil and Bevacizumab
  * Irinotecan (Camtop Injection®, CJ HealthCare Corp.), Leucovorin, 5-Fluorouracil and Cetuximab

SUMMARY:
* Registry
* Multicenter, prospective observational study
* Observe adverse events and efficacy in recruited patients for 3 years under real world settings.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients at least 19 years of age with metastatic colorectal cancer who are planned to receive Bevacizumab or Cetuximab in combination with FOLFIRI regimen as first-line treatment
2. Patients who will receive irinotecan, a component of FOLFIRI regimen, using Camtop Injection®

Exclusion Criteria:

1) Patients with conditions in which any study drug is contraindicated per the respective approved label.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemato oncology clinic
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
percentage of use FOLFIRI regimen and target agents | through study completion, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joong Bae Ahn, Principal Investigator — Severance Hospital, YUHS
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea